CLINICAL TRIAL: NCT01030653
Title: Pharmacokinetics of Voriconazole in Obese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manjunath Prakash Pai (Other)
Collaborators: TKL Research, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Manjunath Prakash Pai, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 09010
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Voriconazole; Pharmacokinetics; Obese; Healthy Volunteer
MeSH Terms: conditions — Obesity | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voriconazole low dose first then high dose (Experimental): Voriconazole administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (200 mg Every 12 Hours x 7 Doses) followed by 7 day washout followed by Loading Dose (400 mg x 2 Doses, Day 1) and a Maintenance Doses (300 mg Every 12 Hours x 7 Doses)
  Interventions: Drug: Voriconazole low dose; Drug: Voriconazole high dose
- Voriconazole high dose first then low dose (Experimental): Voriconazole administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (300 mg Every 12 Hours x 7 Doses) followed by 7 day washout followed by Loading Dose (400 mg x 2 Doses, Day 1) and a Maintenance Doses (200 mg Every 12 Hours x 7 Doses)
  Interventions: Drug: Voriconazole low dose; Drug: Voriconazole high dose

INTERVENTIONS:
Drug: Voriconazole low dose — Voriconazole 400 mg po x 2 doses (loading dose)then 200 mg po twice daily x 7 doses
  Other Names: Vfend
Drug: Voriconazole high dose — Voriconazole 400 mg po x 2 doses (loading dose)then 300 mg po twice daily x 7 doses
  Other Names: Vfend

SUMMARY:
Obese subjects may require a higher fixed oral maintenance dosing regimen of voriconazole compared to normal weight subjects to achieve comparable plasma exposures. The current study is designed to address this issue.

DETAILED DESCRIPTION:
The prevalence of obesity has increased tremendously in the past two decades. An estimated 1 out of 5 persons in the United States are classified as obese. Under representation of obese patients in pharmacokinetic trials grossly limit generalizability of drug dosing recommendations in this emerging population. No published pharmacokinetic studies of voriconazole dosing in patients with obesity currently exist in the literature. Specifically,voriconazole pharmacokinetic data from subjects with a body mass index (BMI) ≥ 35 kg/m2(Class II and III obesity) are limited.

Voriconazole is available as both an intravenous and oral formulation. Anecdotal experience suggest that the use of oral voriconazole to be significantly more prevalent that that of intravenous therapy. The current oral recommended dosing regimen for voriconazole includes use of 200 mg every 12 hours for patients who are over 40 kg. The dosage can be increased to 300 mg by mouth every 12 hours in situations where a sufficient clinical response is not noted. A weight based dosing strategy is also utilized in patients with more serious infections (3-6 mg/kg IV Q 12 hours) such as invasive aspergillosis. Voriconazole demonstrates non-linear pharmacokinetics and so dosing based on total body weight may result in non-dose proportional exposure. For example, a 1.5 fold dose increment in voriconazole from 200 mg to 300 mg every 12 hours results in a 2.5 fold increase in exposure. The most appropriate body size descriptor is unknown (i.e. ideal body weight, fat free weight, lean body weight, etc.) for most antimicrobials, including voriconazole. As a consequence, the appropriateness of weight-based voriconazole dosage selection in obese patients is not known. Intuitively, weight based dosing (on total body weight) in this population could lead to higher than expected exposures (non-linear pharmacokinetics) and lead to potential adverse events. Therapeutic drug monitoring is increasingly advocated as a system to improve voriconazole dosing. However, an assay to measure voriconazole concentrations in the clinic is not routinely available. Hence, the current pilot study proposes to characterize the pharmacokinetic profile of voriconazole in obese subjects using two fixed dose regimens.

ELIGIBILITY:
Inclusion Criteria:

1. males and females, 18 to 50 years of age;
2. non-smoking or light-smoking (≤5 cigarettes per day) volunteers;
3. BMI ≥ 35 kg/m2;
4. female subjects of childbearing potential either surgically sterilized, using an effective method of contraception (diaphragm, cervical cap, condom) or agree to abstain from sex from time of prestudy screening, during entire study period and 1 week following the study period.

Exclusion Criteria:

1. History of significant hypersensitivity reaction or intolerance to voriconazole, fluconazole,itraconazole, posaconazole, or ketoconazole ;
2. history of significant clinical illness requiring pharmacological management;
3. abnormal serum electrolyte or complete blood count requiring further clinical work-up;
4. transaminases (AST or ALT) >2.5 x upper limit of normal;
5. estimated creatinine clearance <50 mL/min (Cockcroft-Gault equation);
6. positive urine pregnancy test (if female);
7. abnormal electrocardiogram (ECG) as judged by study physician;
8. unable to tolerate venipuncture and multiple blood draws;
9. clinically significant abnormal physical examination defined as a physical finding requiring further clinical work-up.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manjunath P Pai, PharmD, Principal Investigator — University of Michigan
Locations (1):
- TKL Research Inc, Paramus, New Jersey, United States

REFERENCES:
- [Background] Pai MP, Norenberg JP, Anderson T, Goade DW, Rodvold KA, Telepak RA, Mercier RC. Influence of morbid obesity on the single-dose pharmacokinetics of daptomycin. Antimicrob Agents Chemother. 2007 Aug;51(8):2741-7. doi: 10.1128/AAC.00059-07. Epub 2007 Jun 4. PMID 17548489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research unit, subjects recruited over a 6 month period
Pre-assignment Details: This was a healthy volunteer study that did not require any pre assignment study procedures. 10 participants were consented but 8 were sufficient to complete the study. The remaining two subjects were not assigned to any arm, comparable to a screen failure. No intervention other than consent and screening occurred for these two subjects.
Groups:
- Voriconazole High Dose First Then Low Dose: Active: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Two Fixed Maintenance Doses ( 300 mg Every 12 Hours x 7 Doses) followed by a 7-day washout period then a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses ( 200 mg Every 12 Hours x 7 Doses)
- Voriconazole Low Dose First Then High Dose: Active: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Two Fixed Maintenance Doses ( 200 mg Every 12 Hours x 7 Doses) followed by a 7-day washout period then a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses ( 300 mg Every 12 Hours x 7 Doses)
Period: Loading Dose & First Maintenance Regimen
Arm/Group | Voriconazole High Dose First Then Low Dose | Voriconazole Low Dose First Then High Dose
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: 7-Day Washout Period
Arm/Group | Voriconazole High Dose First Then Low Dose | Voriconazole Low Dose First Then High Dose
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Loading Dose & 2nd Maintenance Regimen
Arm/Group | Voriconazole High Dose First Then Low Dose | Voriconazole Low Dose First Then High Dose
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Voriconazole High Dose First Then Low Dose: Both voriconazole arms are shown as a single group because the same individuals received both arms of the intervention in a cross-over design.
- Total: Total of all reporting groups
Arm/Group | Voriconazole High Dose First Then Low Dose | Voriconazole Low Dose First Then High Dose | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Steady-State Cmax and Cmin of Two Voriconazole Dosing Regimens
Description: Cmax is the maximum concentration, and Cmin is the minimum concentration. These measurements are based on analysis of plasma. The units shown are milligrams of voriconazole per liter of plasma. The two dosing regimens are:
  1. a loading dose (400 mg x 2 doses, day 1) and maintenance doses (200 mg every 12 hours x 7 doses) in obese subjects.
  2. a loading dose (400 mg x 2 doses, day 1) and maintenance doses (300 mg every 12 hours x 7 doses) in obese subjects.
Time Frame: Day 5
Population: The same subjects were analyzed in a cross-over design at two dose levels
Measure: Mean (95% Confidence Interval); unit: mg/L
Groups:
- Voriconazole Lower Dose: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (200 mg or Every 12 Hours x 7 Doses)
- Voriconazole Higher Dose: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (300 mg or Every 12 Hours x 7 Doses)
Arm/Group | Voriconazole Lower Dose | Voriconazole Higher Dose
Number analyzed (Participants) | 8 | 8
mg/L
  Cmax | 2.36 [1.70 to 3.28] | 4.16 [2.76 to 6.27]
  Cmin | 0.81 [0.46 to 1.44] | 1.76 [1.17 to 2.66]

2. Primary Outcome: Geometric Mean Ratio of the AUC Between the High and Low Dose Voriconazole
Description: AUC is the area under the concentration-time curve. The Geometric Mean Ratio and 90% confidence interval around this value permit an assessment of the bioequivalence of two dosing regimens in the same group. The geometric mean is computed based on the ratio of the AUC value from the high dose compared to the AUC value from the low dose for each individual. This ratio provides a more robust interpretation of the differences between the two dosing arms because each individual serves as their own control.
Time Frame: 14 days
Population: This is a comparison of the same group analyzed through a cross-over design of two voriconazole dosing regimens
Measure: Number (90% Confidence Interval); unit: Ratio
Groups:
- Voriconazole High : Low Dose: 1. Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (200 mg or Every 12 Hours x 7 Doses)
  2. Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (300 mg or Every 12 Hours x 7 Doses)
Arm/Group | Voriconazole High : Low Dose
Number analyzed (Participants) | 8
Ratio | 2 [1.5 to 2.7]

3. Secondary Outcome: The Area Under the Curve Over the Dosing Interval for All Participants While on the High Dose and Low Dose Interventions.
Time Frame: 12 hours
Measure: Geometric Mean (95% Confidence Interval); unit: hour*milligram/Liter
Arm/Group | Voriconazole Lower Dose | Voriconazole Higher Dose
Number analyzed (Participants) | 8 | 8
hour*milligram/Liter | 14.6 [9.21 to 23.1] | 29.2 [19.4 to 43.8]

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Voriconazole High Dose: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (300 mg or Every 12 Hours x 7 Doses)
- Voriconazole Low Dose: Voriconazole Administered by Mouth as a Loading Dose (400 mg x 2 Doses, Day 1) and as Maintenance Doses (200 mg or Every 12 Hours x 7 Doses)
Arm/Group | Voriconazole High Dose | Voriconazole Low Dose
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The study sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No